CLINICAL TRIAL: NCT03994575
Title: North American Acute Coronary Syndrome (ACS) Reflective III Pilot
Status: Completed | Type: Observational
Sponsor: Canadian Heart Research Centre (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Dr. Anatoly Langer, Director, Canadian Heart Research Centre
Other Study IDs: DCV-2017-11935
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Dyslipidemias; Acute Coronary Syndrome
MeSH Terms: conditions — Dyslipidemias; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Guideline recommended feedback — The ACS Reflective III Pilot program is a quality assurance program where the decision to follow the recommendations and all treatment decisions related to patient care are left to the physician's discretion and feedback to the physician with their aggregate and individual patient data is intended as a quality assurance undertaking

SUMMARY:
The North American ACS Reflective III Pilot is an observational, Quality Enhancement Research Initiative (QuERI), knowledge translation program designed to give feedback to physicians on their post-ACS lipid-lowering management in an effort to support their decision-making and choice of therapies and thereby better achieve evidence-based, guideline-recommended management of post-ACS patients. The ACS Reflective III Pilot follows the completed ACS Registries I, II, and III, ACS Reflective I, and the ongoing ACS Reflective II programs.

DETAILED DESCRIPTION:
The main objectives are:

1. To identify and describe post-ACS patients who do not achieve guideline-recommended LDL-C "target" (<1.8 mmol/L in Canada, >50% LDL-C lowering on high-intensity statin in the U.S.);
2. To identify opportunities where PCSK9 inhibitor therapy may be of potential benefit in the management of post-ACS patients to achieve guideline-recommended LDL-C goal by 1 year follow-up; and,
3. To determine reasons why physicians are not prescribing guideline-recommended LDL-C lowering therapies and/or patients are not achieving guideline-recommended LDL-C goals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age;
2. ACS 1-12 months prior to enrolment defined by symptoms of myocardial ischemia with an unstable pattern, occurring at rest or with minimal exertion, within 72 hours of an unscheduled hospital admission due to presumed or proven obstructive coronary disease and at least one of the following:

   1. Elevated cardiac biomarkers (e.g., troponin) = myocardial infarction (MI); or,
   2. Resting ECG changes consistent with ischemia, plus additional evidence of obstructive coronary disease from regional wall motion or perfusion abnormality, 70% or greater epicardial coronary stenosis by angiography, or need for coronary revascularization procedure = unstable angina (UA); and,
3. LDL-C ≥1.81 mmol/L (70 mg/dL) despite maximally tolerated statin ± ezetimibe therapy (including patients who are intolerant of ≥2 statins).

Exclusion Criteria:

1. Participating in a research study where the lipid-modifying therapy is unknown, randomly assigned (i.e., choice not determined by the physician), or not approved for clinical use; or
2. Follow-up or life expectancy <1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 years or older, 1-12 months post-ACS, with LDL-C ≥1.81 mmol/L (70 mg/dL) despite maximally tolerated statin ± ezetimibe therapy (including patients who are intolerant of ≥2 statins).
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving Canadian and American guideline-recommended LDL-cholesterol goal(s) | 12 months
  The primary endpoint is the proportion of patients achieving Canadian and American guideline-recommended goals (i.e., LDL-C ≤1.8 mmol/L [70 mg/dL] or >50% LDL-C reduction, respectively, after the final visit (Visit 3; approximately 1 year post-ACS). (If, during the course of the study, the guideline-recommended LDL-C goal changes, both the current and new goals will be considered).

SECONDARY OUTCOMES:
Relative reduction of LDL-C achieved | 3-6 and 6-12 months, respectively
Proportion of patients achieving guideline-recommended targets | 3-6 months
Proportion of patients receiving additional lipid-modifying therapies (including PCSK9 inhibition) | 3-6 and 6-12 months, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Shaun G Goodman, MD, MSc, Principal Investigator — Co-Chair, Canadian Heart Research Centre
Locations (1):
- Canadian Heart Research Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No